CLINICAL TRIAL: NCT02474823
Title: Neck Grasp as a Predictor of Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, Lee Edmonds, MD, attending physician - Pulmonology, Bassett Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012
Record Dates: First submitted 2015-06-09; First posted 2015-06-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Obstructive Sleep Apnea; Type 2 Diabetes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep Apnea assessment (Other): all participants are in the same arm & undergo the same assessments: PSG, HST, ESAP
  Interventions: Other: polysomnogram; Other: home sleep test; Other: Easy Sleep Apnea Predictor

INTERVENTIONS:
Other: polysomnogram — all participants will undergo PSG for assessment of OSA
  Other Names: PSG
Other: home sleep test — all participants will undergo HST for assessment of OSA
  Other Names: HST
Other: Easy Sleep Apnea Predictor — all participants will undergo ESAP for assessment of OSA
  Other Names: ESAP , self neck grasp

SUMMARY:
A previous pilot study on the use of self neck grasp, ESAP (Easy Sleep Apnea Predictor), showed a positive maneuver (unable to wrap hands completely around neck) to be 100% predictive of sleep apnea in a sleep clinic population. The investigators now would like to compare ESAP to other tests used to diagnose and screen for Sleep Apnea in type 2 diabetics. The tests will included Home Sleep Testing, sleep questionnaires Berlin and STOP-BANG and polysomnogram (PSG). Patients with type 2 diabetes in the Bassett Endocrine Clinic who are scheduled for a routine evaluation will be recruited to undergo; a Home Sleep Test along with two sleep questionnaires PSG. The screen test wil be compared to the results of the gold standard diagnostic test the PSG for their predictive value os OSA in the type 2 diabetic population.

DETAILED DESCRIPTION:
The goal is to evaluate the ESAP study (simple neck grasp) as a predictor of Obstructive Sleep Apnea (OSA) in combination with, and in comparison to; Home Sleep Test ( HST), Berlin Sleep Questionnaire and STOP-BANG questionnaire. All predictors are being evaluated against the gold standard test, the polysomnogram (PSG).

OSA is the common disorder affecting 3-7% of the adult population. It has many negative health consequences such as; cardiovascular disease, diabetes, motor vehicle accidents and depression. Data from both epidemiological and clinical studies suggest that OSA is also independently associated with alterations in glucose metabolism and places patients at an increased risk of the development of type 2 diabetes It is often missed in a busy practice. This simple diagnostic tool may help us in identifying the patient at an earlier stage, thus also helping to prevent further complications in diabetic patients.

Participants will undergo 3 study visits/procedures:

Visit 1: Participants will be consented for the study, undergo the ESAP test, complete the Berlin Sleep Questionnaire & STOP-BANG questionnaire, and provide medical history/demographic information.

Visit 2: Participants will undergo a PSG at the Bassett Sleep Lab.. Visit 3: The morning the PSG is completed, participants will be given the HST recorder and instructed in its use in order to complete the HST. Participants can then drop off the HST recorder at any Bassett Clinic and it will be returned to the Sleep Lab in Cooperstown.

The ESAP test, Berlin Sleep Questionnaire, and the STOP-BANG Questionnaire will be administered by a study coordinator, research nurse, and/or research assistant. The PSG and the HST will be read and evaluated by independent evaluators/physicians. These physicians will not have access to the ESAP or the questionnaire results prior to the evaluation of the PSG or HST.

If a participant has any test (except the ESAP test alone) that is indicative or suspicious for OSA, a study physician will review these results and advise them of any further follow up recommendations.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years old regardless of gender
* Confirmed diagnosis of Type 2 diabetes

Exclusion Criteria:

* Unstable Heart failure
* COPD
* Neuromuscular disease
* Mental disorders which would interfere with following directions
* Persons who are already diagnosed with OSA or persons who have been using CPAP or BiPAP

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Result of ESAP testing | 3 months
  The ESAP measures a participant's ability to wrap their own hands around their neck, touching thumb to thumb, middle finger to middle finger. A "positive" test (unable to reach around the neck with fingers) would be indicative of the presence of OSA.

SECONDARY OUTCOMES:
results of HST | 3 months
  Positive HST would indicate presence of OSA
Result of PSG testing | 3 months
  Positive PSG would indicate presence of OSA

CONTACTS AND LOCATIONS:
Overall Officials: lee edmonds, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

REFERENCES:
- [Derived] Edmonds PJ, Gunasekaran K, Edmonds LC. Neck Grasp Predicts Obstructive Sleep Apnea in Type 2 Diabetes Mellitus. Sleep Disord. 2019 Jul 1;2019:3184382. doi: 10.1155/2019/3184382. eCollection 2019. PMID 31355009